CLINICAL TRIAL: NCT06408922
Title: Comparison of the Effects of Single Versus Triple Injections of Platelet-Rich Plasma in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: prpknee2023
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Pituitary Adenylate Cyclase-Activating Polypeptide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single prp injection (Active Comparator): single intraarticular prp injection
  Interventions: Other: prp injection
- triple prp injection (Active Comparator): triple intraarticular prp injection
  Interventions: Other: prp injection

INTERVENTIONS:
Other: prp injection — intraarticular prp

SUMMARY:
80 patients diagnosed with knee osteoarthritis were randomized into two groups: patients in Group 1 received a single intraarticular injection of PRP whereas those in group 2 were administered three intraarticular injections of PRP within an interval of 2 weeks between each application. Patients were evaluated before the treatment and at the 6 month after the treatment with a Visual Analog Scale (VAS) and The Western Ontario and MacMaster Universities (WOMAC) Osteoarthritis Index.

ELIGIBILITY:
Inclusion Criteria:

* ages of 35 and 80
* Kellgren-Lawrence grade of 2, 3, or 4

Exclusion Criteria:

* rheumatic diseases, coagulopathies, severe cardiovascular diseases, local infections, malignancies, immunodeficiency, schizophrenia, mental retardation, anticoagulant therapy, a hemoglobin concentration of 11 g/dL and platelets of 150,000/L, a history of severe trauma, or a history of hyaluronic acid or corticosteroid injection within the previous 6 months

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
The Western Ontario and MacMaster Universities (WOMAC) Osteoarthritis Index | baseline and 6 months

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | baseline and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Buca Seyfi Demirsoy Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No